CLINICAL TRIAL: NCT00027885
Title: A Randomized Phase II Study of Bevacizumab in Combination With Docetaxel in Locally Advanced Breast Cancer
Brief Title: Phase II Bevacizumab + Tax In Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CWRU3100; U01CA062502 (NIH); P30CA043703 (NIH); CWRU-3100 (Other: Case Comprehensive Cancer Center); NCI-2722 (Other: CTEP/NCI)
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Bevacizumab; Cyclophosphamide; Docetaxel; Doxorubicin; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docetaxel (Active Comparator): Patients receive docetaxel IV over 1 hour once weekly on weeks 1-6.
  Interventions: Drug: cyclophosphamide; Drug: docetaxel; Drug: doxorubicin hydrochloride; Procedure: adjuvant therapy; Procedure: conventional surgery; Procedure: neoadjuvant therapy; Radiation: radiation therapy
- Combine bevacizumab and docetaxel. (Experimental): Patients receive docetaxel IV over 1 hour once weekly on weeks 1-6 and bevacizumab IV over 60 minutes once every 2 weeks on weeks 1-8.
  Interventions: Biological: bevacizumab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Procedure: adjuvant therapy; Procedure: conventional surgery; Procedure: neoadjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Biological: bevacizumab — Patients receive bevacizumab IV over 60 minutes once every 2 weeks on weeks 1-8.
  Arms: Combine bevacizumab and docetaxel.
Drug: cyclophosphamide — Approximately 4 weeks after the completion of radiotherapy, patients receive cyclophosphamide IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
Drug: docetaxel — Patients receive docetaxel IV over 1 hour once weekly on weeks 1-6.
  Other Names: Taxotere
  Arms: Docetaxel
Drug: doxorubicin hydrochloride — Approximately 4 weeks after the completion of radiotherapy, patients receive doxorubicin IV over 5 minutes. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
Procedure: adjuvant therapy — After the second course, patients with stable or responsive disease undergo modified radical mastectomy or breast-conserving surgery. Three to six weeks after surgery, patients undergo radiotherapy 5 days a week for 7 weeks.
  Approximately 4 weeks after the completion of radiotherapy, patients receive doxorubicin IV over 5 minutes and cyclophosphamide IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
Procedure: conventional surgery — After the second course, patients with stable or responsive disease undergo modified radical mastectomy or breast-conserving surgery.
Procedure: neoadjuvant therapy — Arm I: Patients receive docetaxel IV over 1 hour once weekly on weeks 1-6 and bevacizumab IV over 60 minutes once every 2 weeks on weeks 1-8.
  Arm II: Patients receive docetaxel as in arm I. Treatment in both arms repeats every 8 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.
Radiation: radiation therapy — Three to six weeks after surgery, patients undergo radiotherapy 5 days a week for 7 weeks.

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or deliver cancer-killing substances to them. Combining chemotherapy with monoclonal antibody therapy may kill more tumor cells.

PURPOSE: This randomized phase II trial is to see if docetaxel with or without bevacizumab followed by surgery, radiation therapy, and combination chemotherapy works better in treating patients who have stage III or stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of bevacizumab and docetaxel on reduction of microvessel density and induction of apoptosis of endothelial and tumor cells in patients with locally advanced breast cancer.
* Determine the safety profile of this regimen in these patients.
* Compare the effect of docetaxel and bevacizumab, in terms of objective response, stabilization of disease, and progression-free survival, in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to disease stage. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive docetaxel IV over 1 hour once weekly on weeks 1-6 and bevacizumab IV over 60 minutes once every 2 weeks on weeks 1-8.
* Arm II: Patients receive docetaxel as in arm I. Treatment in both arms repeats every 8 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.

After the second course, patients with stable or responsive disease undergo modified radical mastectomy or breast-conserving surgery. Three to six weeks after surgery, patients undergo radiotherapy 5 days a week for 7 weeks.

Approximately 4 weeks after the completion of radiotherapy, patients receive doxorubicin IV over 5 minutes and cyclophosphamide IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients with estrogen and/or progesterone receptor-positive disease also receive oral tamoxifen daily for 5 years beginning after the completion of chemotherapy. Post-menopausal patients may receive oral anastrozole once daily for 5 years instead of tamoxifen.

Patients are followed at 3, 6, and 12 months, every 6 months for 4 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 60 patients (30 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast

  * Stage IIIA or IIIB
  * Stage IV if patient has clinical evidence of locally advanced breast cancer only
  * Inoperable disease
* Prior carcinoma in situ of the breast or bilateral breast cancer is allowed
* No CNS metastases
* Hormone receptor status:

  * Estrogen and progesterone receptor status known

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female or male

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy:

* More than 6 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal (no greater than 2 times upper limit of normal [ULN] in patients with an inherited disorder)
* AST/ALT no greater than 2.5 times ULN
* INR and PTT normal

Renal:

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min
* No proteinuria or clinically significant renal impairment

Cardiovascular:

* LVEF at least 45% by echocardiogram or MUGA scan
* No New York Heart Association class III or IV heart disease
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No inadequately controlled hypertension
* No history of deep vein thrombosis or other thromboses
* No clinically significant peripheral artery disease
* No arterial thromboembolic event within the past 6 months including the following:

  * Transient ischemic attack
  * Cerebrovascular accident
  * Myocardial infarction

Other:

* No other prior or concurrent malignancy within the past 10 years except inactive nonmelanoma skin cancer or carcinoma in situ of the cervix
* No other uncontrolled concurrent illness
* No ongoing or active infection
* No non-healing wounds
* No psychiatric illness or social situation that would preclude study participation
* No prior allergic reaction to compounds of similar chemical or biological composition to bevacizumab, docetaxel, polysorbate 80 (Tween) formulations, or other agents used in this study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent cytokines during docetaxel/bevacizumab administration

  * Concurrent cytokines during doxorubicin/cyclophosphamide administration allowed at the discretion of the treating physician

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Prior hormonal therapy (e.g., tamoxifen) allowed

Radiotherapy:

* Prior radiotherapy to affected breast allowed

Surgery:

* More than 28 days since prior major surgery

Other:

* At least 10 days since prior thrombolytic agents
* At least 10 days since prior full-dose oral or parenteral anticoagulants except to maintain patency of permanent indwelling IV catheters
* Concurrent warfarin allowed provided INR is less than 1.5
* Concurrent bisphosphonates allowed for osseous metastases provided they are not initiated on day 1 of cycle 1
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent full-dose oral or parenteral anticoagulants except to maintain patency of permanent indwelling IV catheters
* No concurrent thrombolytic agents
* No other concurrent anticancer agents or therapies
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2001-11; Primary Completion 2005-12 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the ability of bevacizumab and docetaxel to reduce microvessel density and induce apoptosis of endothelial and tumor cells. | weeks 8 and 17
  The primary outcome measure is the difference in change in biologic parameters between the two arms. Tumor biopsies are required to perform pre- and post-treatment tumor microvessel density determination, apoptosis by TUNEL assay, proliferation markers by immunohistochemistry(e.g. PCNA, Ki-67), and expression of nuclear clusterin/XIP8.

SECONDARY OUTCOMES:
Number of patients with objective response | 5 years
  Response and progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee

CONTACTS AND LOCATIONS:
Overall Officials: Paula Silverman, MD, Study Chair — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (5):
- United States (5):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - UH-Southwest, Middleburg Heights, Ohio
  - UH-Chagrin Highlands, Orange, Ohio
  - UH-Green Road, South Euclid, Ohio
  - UH-Westlake, Westlake, Ohio